CLINICAL TRIAL: NCT04860817
Title: Investigating the Safety and Efficacy of Anti-CD7 CAR-T Cell Immunotherapy in Patients With Relapse and Refractory T-cell Acute Lymphoblastic Leukemia or T Lymphoblastic Lymphoma
Brief Title: A Study of Anti-CD7 CAR-T Cells in Pediatric and Young Adult Patients With Relapse and Refractory T-ALL/ T-LBL
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No proper participant is found.
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUT03
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-lymphoblastic Lymphoma
Keywords: CAR-T; CD7; T-ALL/LBL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target CD7 CAR-T cells (Experimental): Three dose levels will be evaluated. The CAR-T cells will be administered with Cytoxan and fludarabine.
  Interventions: Biological: Target CD7 CAR-T cells

INTERVENTIONS:
Biological: Target CD7 CAR-T cells — Enrolled participants are allocated to one of three different dose levels of target CD7 CAR-T cells. The infusion dose of CAR-T cells will start at low dose and then rise to higher dose after completion of low dose group.
  1. Dose level one: 0.6×10^7 cells/kg;
  2. Dose level two: 1×10^7 cells/kg;
  3. Dose level three: 1.5×10^7 cells/kg. Before CAR-T infusion, all participants will receive a preconditioning therapy suggested as: Fludarabine 30 mg/m^2×6d, Cyclophosphamide 300 mg/m^2×6d or Cyclophosphamide 600 mg/m^2×6d. After completion of preconditioning therapy, infusion of CAR-T cells needs to start within 1 week. Participants will receive one infusion of CAR-T cells which will take between 15 and 30 mins.

SUMMARY:
T cells are a type of immune cell. Like other cells of the body, T Cells can develop cancer. T cell cancers mainly include T cell leukaemia and T cell lymphoma, both of which have a relatively poor prognosis. Currently, patients with relapsed/refractory type (the name given to cancer that reappears or grows again after a period of no changes or signs of cancer) of this leukaemia or lymphoma have limited choices for treatment. CAR-T cells are immune cells that are engineered to target specific cell markers. For example, CAR-T cells targeting the marker CD19 have shown great effectiveness in the treatment of B cell tumors that carry this marker. Here investigators construct a new universal CAR-T design targeting CD7 which is found on the cells of relapsed/refractory type T cell leukaemia and lymphoma and hope to test its safety and efficiency in the treatment of relapsed/refractory type T cell leukaemia and lymphoma.

DETAILED DESCRIPTION:
Who can participate? Patients diagnosed with relapsed/refractory T cell leukaemia or lymphoma. Both genders, aged 2-25 years old.

What does the study involve? Enrolled participants are randomly chosen to receive one of three different dose levels of CAR-T cells.

1. Dose level one: 0.6×10^7 cells/kg;
2. Dose level two: 1×10^7 cells/kg;
3. Dose level three: 1.5×10^7 cells/kg. Before CAR-T infusion, all participants will receive a preconditioning therapy including several chemotherapy agents or other interventions that are required to help the effect of the CAR-T cells. After completion of preconditioning therapy, infusion of the CAR-T cells via a tube into the vein needs to start within 1 week. Participants will receive one infusion of CAR-T cells which will take between 15 and 30 mins. All participants will have a blood test before infusion and at 4, 7, 10 and 14 days following infusion to measure their response to the treatment and some further tests will be required in some participants.

What are the possible benefits and risks of participating? The universal CAR-T cells targeting CD7 may lead to durable disease control and long term survival. The main risks of participating include cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS).

Where is the study run from? Haematology department of 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (China).

ELIGIBILITY:
Inclusion Criteria:

1. 2 to 25 years
2. Diagnosed with relapsed and refractory CD7 + T cell acute lymphocytic leukemia (T-ALL) or relapsed and refractory CD7 + T lymphoblastic lymphoma (T-LBL)
3. Quantifiable tumor burden
4. Eastern cooperative oncology group (ECOG) performance status of 0 to 1
5. Life expectancy ≥12 weeks
6. Adequate organ function defined as:

   1. Serum ALT/AST ≤2.5 ULN
   2. Creatinine clearance (as estimated by Cockcroft Gault) ≥60 mL/min
   3. PT and APTT≤1.5 ULN
   4. Total bilirubin ≤1.5 ULN
   5. Cardiac ejection fraction ≥45%
   6. No clinically significant ECG findings
   7. Baseline oxygen saturation >90% on room air
7. Recovered from acute toxic effects of prior chemotherapy ≥one week before entering this study
8. Agreement to use of medical-approved-contraception during the period of trial and in 1 year after cell transfusion therapy
9. Signed informed consent form

Exclusion Criteria:

1. Diagnosis of other malignancy (except non-melanoma and cervical carcinoma in situ, bladder cancer, breast cancer that have a disease-free survival of more than 5 years)
2. Severe mental disorders
3. History of hereditary diseases, including but not limited to: Fanconi anemia, Shut-Dai syndrome, Costman syndrome or any other known bone marrow failure syndrome
4. Grade 2-4 acute graft-versus-host disease (GVHD) (Glucksberg criteria) or extensive chronic GVHD (Seattle criteria)
5. Grade III-IV heart failure or myocardial infarction, angioplasty or stent placement, unstable angina pectoris, or other clinically prominent heart disease within one year before enrollment
6. History or presence of CNS disorder, including but not limited to: seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
7. Positive for any of the following etiological tests: HIV, HBV, HCV, TPPA
8. Presence of fungal, bacterial, viral, or other infection that is uncontrolled
9. Severe allergies
10. History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
11. History or diagnosis of pulmonary fibrosis
12. Participation in other clinical trials ≤4 weeks prior to enrollment
13. Concomitant disease that require systemic steroids or other immune suppressive therapy during the study period in researcher's judgement
14. Patients who are contraindicated to cyclophosphamide, fludarabine
15. Allogeneic cell therapy (such as donor lymphocyte infusion, DLI) ≤6 weeks prior to enrollment
16. Poor adherence due to physical, family, social, geographic, and other factors, who cannot follow the research plan and follow-up plan
17. Pregnant and lactating women
18. Any other conditions that researcher think it is inappropriate for the subject to anticipate the trial

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity | up to 4 weeks after target CD7 CAR-T cells infusion
  Dose-limiting toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0) at 4 weeks following target CD7 CAR-T cells infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | 4 weeks, 12 weeks, 24 weeks after target CD7 CAR-T cells infusion
  ORR of patients, determined by National Comprehensive Cancer Network (NCCN) clinical practice guidelines in oncology: Acute Lymphoblastic Leukemia (2016.V2) for T-ALL response rate and Lugano 2014 for T-LBL response rate.
Progression-free survival (PFS) | 24 weeks after target CD7 CAR-T cells infusion
  PFS determined from patient notes at 24 weeks following target CD7 CAR-T cells infusion.
Overall survival (OS) | 24 weeks after target CD7 CAR-T cells infusion
  OS determined from patient notes at 24 weeks.
Duration of remission (DOR) | 24 weeks after target CD7 CAR-T cells infusion
  DOR determined from patient notes at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No